CLINICAL TRIAL: NCT04521296
Title: A Double-blind, Randomized, Placebo-controlled, Multi-center, Phase II/III Study to Evaluate the Efficacy and Safety of DWJ1248 in Patients With Mild to Moderate COVID-19
Brief Title: Efficacy and Safety of DWJ1248 in Patients With Mild to Moderate COVID-19 Compared to the Placebo
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Changes in drug development plans
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1248201
Record Dates: First submitted 2020-07-07; First posted 2020-08-20 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2021-10

CONDITIONS: Mild to Moderate COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWJ1248 (Experimental): Camostat mesylate
  Interventions: Other: Part 1; Other: Part 2
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Part 1; Other: Part 2

INTERVENTIONS:
Other: Part 1 — - DWJ1248 600mg PO (100mg 2 tab, TID)
Other: Part 2 — - DWJ1248 600mg PO (200mg 1 tab, TID)

SUMMARY:
To evaluate the efficacy and safety after administration of DWJ1248 in patients with mild to moderate COVID-19 compared to the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 19 as of the signed date in written consent
* Subjects with mild or moderate COVID-19 according to RT-PCR test (Total score of NEWS is 0-6 or if one item is 3 points)
* Subjects who have symptoms within 7 days or 72 hours after diagnosis

Exclusion Criteria:

* Subjects who cannot orally administer the investigational products
* Subjects who need administration of immunosuppressants
* Subjects who are allergic or sensitive to investigational products or its ingredients
* Subjects who have a history of drug and/or alcohol abuse within 52 weeks before screening
* Subjects who have been identified with uncontrolled concomitant diseases or conditions, including significant mental illness and social conditions, that may affect compliance with clinical trial procedures according to the determination of the investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
(Part 1) Time to SARS-CoV-2 eradication | Up to 28 days
  Time to reach undetectable SARS-CoV-2 RNA level
(Part 2) Time to clinical improvement of subjective symptoms | Up to 14 days
  Clinical improvement of subjective symptoms (days)

SECONDARY OUTCOMES:
(Part 1) Rate of SARS-CoV-2 eradication | Days 4, 7, 10, and 14
  Percent of patients with undetectable SARS-CoV-2 RNA level
(Part 1/2) Time to clinical improvement of subjective symptoms | Up to 28 days
(Part 2) Change from baseline of subjective symptom scores | Days 4, 7, 10, 14, 21 and 28

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim YS, Jeon SH, Kim J, Koh JH, Ra SW, Kim JW, Kim Y, Kim CK, Shin YC, Kang BD, Kang SJ, Park CH, Lee B, Lee JY, Lee CH, Choi JP, Kim JY, Yu SN, Peck KR, Kim SH, Heo JY, Kim HA, Park HJ, Choi J, Han J, Kim J, Kim HJ, Han SH, Yoon A, Park M, Park S, Kim Y, Jung M, Oh MD. A Double-Blind, Randomized, Placebo-Controlled, Phase II Clinical Study To Evaluate the Efficacy and Safety of Camostat Mesylate (DWJ1248) in Adult Patients with Mild to Moderate COVID-19. Antimicrob Agents Chemother. 2023 Jan 24;67(1):e0045222. doi: 10.1128/aac.00452-22. Epub 2022 Dec 14. PMID 36515544